CLINICAL TRIAL: NCT06810674
Title: Get Out of Your Head 2.0: Evaluation of an Online Prevention Campaign and Updated Website for Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0537
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Suicide; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Get Out of your head campaign and website 2.0 (Experimental): Participants in this group (all participants) are asked to complete a questionnaire (15-20 min). After completing these measures, participants will view the developed campaign materials (visuals) and will be asked to provide feedback. Subsequently, participants will receive a link to the website, along with instructions to review the new content pages. They will have three days to explore the site before receiving an email prompting them to complete the post-test questionnaire (10-15 min), which will take approximately 10-15 minutes. If the post-test is not completed after seven or eight days, a reminder will be sent.
  Interventions: Behavioral: Get out of your head campaign and website 2.0

INTERVENTIONS:
Behavioral: Get out of your head campaign and website 2.0 — The Get out of your head campaign and website were launched in 2022 to improve men's mental health and reduce stigma (Stas et al., 2024). Developed with experts, a communication agency, and the target audience, the campaign included videos, testimonies, and a website with tailored information on mental health, suicide prevention, and help-seeking (www.komuitjekop.be).
  The new campaign and updated website will focus specifically on facilitating help-seeking behaviour among men experiencing suicidal thoughts by increasing their perceived need for support. More specifically, the new campaign will aim to enhance the recognition of their suffering, the relevance of seeking and receiving help and changing the perception of suicidal thoughts, namely that these are not fixed or part of life, but instead are changeable and can improve with the correct help.

SUMMARY:
The primary objective of this study is to evaluate the perceptions and evaluations of men with suicidal thoughts, regarding the new "Get Out of Your Head" campaign and the updated website. The findings will inform potential adjustments to enhance the campaign and website as needed.

DETAILED DESCRIPTION:
In a previous study (BUN: B6702024000090) the authors focused on identifying these barriers and needs among adult men experiencing suicidal thoughts and their healthcare providers. Findings from this needs assessment suggest that men with suicidal ideation often perceive a lower need for help and hold attitudes that inhibit help-seeking and sustained engagement in care. These attitudes appear closely linked to societal gender norms around emotional openness, self-reliance, and the perceived responsibility to provide for a family. Furthermore, men experiencing suicidal thoughts expressed a desire for information on certain topics that may currently be unavailable.

To address these gaps, a new awareness campaign is being developed, alongside updates to the existing "Get out of your head" website (original: www.komuitjekop.be), incorporating necessary information. The campaign and website updates are being shaped through a participatory co-creation process involving men with a history of suicidal thoughts to ensure relevance and leverage their experiential knowledge (BUN: B6702024000420). In this approach, men with lived experience are central to the decisions on the design and content of the tools. Additionally, input from experts in healthcare and masculinity, as well as international research, is being integrated.

Once the campaign is developed and the website (www.komuitjekop.be) is updated, the authors aim to evaluate how these resources are perceived by men with suicidal thoughts to further refine these suicide prevention efforts.

The primary objective of the current study is to evaluate the perceptions and evaluations of men with suicidal thoughts, regarding the new "Get Out of Your Head" campaign and the updated website. The findings will inform potential adjustments to enhance the campaign and website as needed.

ELIGIBILITY:
Inclusion Criteria:

* Men (≥ 18y/o)
* Experienced suicidal thoughts in the past three year
* Access to a smartphone, tablet, or computer with internet connection
* Proficiency in Dutch

Exclusion Criteria:

* Does not meet the specified inclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Experienced need | Change from Baseline (before intervention) to post-test (after viewing campaign during 3days); time frame of 3 days
  1 Question based on previous study : to what extent they feel they need support or help from others, on a scale of 0 (not at all) to 10 (a lot), with higher scores indicating a higher perceived need

SECONDARY OUTCOMES:
Attitudes about suicidal thoughts and help-seeking | Change from Baseline (before intervention) to post-test (after viewing campaign during 3days); time frame of 3 days
  5 items from the Attitudes Towards Suicide (ATTS); 3 adapted items from the Attitudes Toward Seeking Professional Psychological Help Scale (ATSPPHS); 4 items from the Network Orientation Scale. All items (12) are to be rated on a scale of 1 (totally disagree) to 5 (totally agree), resulting in a score between 12 and 60.
Help-seeking intention | Change from Baseline (before intervention) to post-test (after viewing campaign during 3days); time frame of 3 days
  Shortened version of the General Helpseeking Questionnaire: 7 items (Healthcare provider; helpline, general practitioner, psychiatrist, close one, other, no one) to be rated on a scale from 1 (extremely unlikely) to 7 (extremely likely) of how likely they are to ask those people for help. Higher scores indicate a higher intention to seek help. Range: 7-49.
Evaluation of the campaign materials | Baseline
  Evaluation statements and open questions for feedback: would they visit the website (yes/no), which information would they expect on the website (open question); 10 statements to be rated on a scale of 1 (totally disagree) to 5 (totally agree); 3 open questions for feedback
Evaluation of the new/updated webcontent | Post-test (after viewing campaign), assessed 3 days after pretest
  Evaluation statements and open questions for feedback: 9 statements to be rated on a scale of 1 (totally disagree) to 5 (totally agree); 3 open questions for feedback.

OTHER OUTCOMES:
Socio-demographic characteristics | Baseline
  self-developed questionnaire: Age, relationship status, work status, education, ethnicity, province, Familiar with 'get out of your head' campaign
Suicidality | Baseline
  Suicidal thoughts and behavior based on questions from the national health survey: suicidal ideation ever (no; yes once; yes more than once); suicidal ideation past year (yes/no); suicide attempt ever (no; yes once; yes more than once); suicide attempt past year (yes, no)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — Flemish Centre of Expertise in Suicide Prevention (Ghent University)
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanlon CA, Chopra J, Boland J, McIlroy D, Poole H, Saini P. A mixed-methods evaluation of the acceptability and fidelity of the James' Place model for men experiencing suicidal crisis. Health Psychol Behav Med. 2023 Oct 11;11(1):2265142. doi: 10.1080/21642850.2023.2265142. eCollection 2023. PMID 37842012
- [Background] Boyle, E. (2007),
- [Background] Watling D, Preece M, Hawgood J, Bloomfield S, Kolves K. Developing an Intervention for Suicide Prevention: A Rapid Review of Lived Experience Involvement. Arch Suicide Res. 2022 Apr-Jun;26(2):465-480. doi: 10.1080/13811118.2020.1833799. Epub 2020 Oct 18. PMID 33073734
- [Background] Stas P, De Jaegere E, van Heeringen K, Ballon A, Portzky G. Evaluation of an online suicide prevention campaign targeting men. Suicide Life Threat Behav. 2024 Feb;54(1):95-107. doi: 10.1111/sltb.13021. Epub 2023 Nov 16. PMID 37970735
- [Background] Renberg ES, Jacobsson L. Development of a questionnaire on attitudes towards suicide (ATTS) and its application in a Swedish population. Suicide Life Threat Behav. 2003 Spring;33(1):52-64. doi: 10.1521/suli.33.1.52.22784. PMID 12710540
- [Background] Mackenzie, C. S., Knox, V. J., Gekoski, W. L., & Macaulay, H. L. (2004). An Adaptation and Extension of the Attitudes Toward Seeking Professional Psychological Help Scale. Journal of Applied Social Psychology, 34(11), 2410-2435. https://doi.org/10.1111/j.1559-1816.2004.tb01984.x
- [Background] Fischer, E. H., Farina, A. (1995). Attitudes toward seeking professional psychological help: A shortened form and considerations for research. Journal of College Student Development, 36, 368-373.
- [Background] Vaux, A. (1985). Factor Structure of the Network Orientation Scale. Psychological Reports, 57(3_suppl), 1181-1182. https://doi.org/10.2466/pr0.1985.57.3f.1181
- [Background] Wilson, C. J., Deane, F. P., Ciarrochi, J. V., & Rickwood, D. (2005). Measuring help seeking intentions: properties of the general help seeking questionnaire.
- [Background] Tang S, Reily NM, Arena AF, Batterham PJ, Calear AL, Carter GL, Mackinnon AJ, Christensen H. People Who Die by Suicide Without Receiving Mental Health Services: A Systematic Review. Front Public Health. 2022 Jan 18;9:736948. doi: 10.3389/fpubh.2021.736948. eCollection 2021. PMID 35118036
- [Background] Gisle, L., Drieskens, S., Demarest, S., & van der Heyden, J. (2020). Geestelijke gezondheid: Gezondheidsenquête 2018. www.gezondheidsenquete.be